CLINICAL TRIAL: NCT05968872
Title: Assessing Knowledge and Attitude of Health Professionals Towards Anesthesia and Anesthetist's Role in the Health Delivery System at Dessie Comprehensive Specialized Hospital, From May 1st to September 30th, 2022, G.C.
Brief Title: Assessing Knowledge & Attitude of Health Professionals Towards Anesthesia and the Anesthetist's Role.
Status: Completed | Type: Observational
Sponsor: Wollo University (Other)
Responsible Party: Principal Investigator, Aynalem Befkadu Woldemichael, Lecturer, Wollo University
Other Study IDs: 6525
Record Dates: First submitted 2023-05-13; First posted 2023-08-01 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Knowledge; Attitude
Keywords: Anesthesia; Attitude; Ethiopia; Health profetionals; knowledge
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: no intervation — it is observational, no intervention was taken

SUMMARY:
Misconceptions about anesthesia and anesthetists in the health professional community may limit anesthetists' participation in their roles. These misconceptions affect the morals of anesthetists since their activity will be limited only to operation theater and the community at large, who did not get the desired care. Improving health professionals' awareness of anesthesia will make it easier for anesthetists to practice their full role and to develop a sense of validation by having their importance acknowledged. Moreover, society will gate the care offered by the anesthetist in different places of medical care.

DETAILED DESCRIPTION:
Data were collected using self-administered, pretested questionnaires prepared in english and then translated into amharic. The Amharic version of the questionnaire was assessed for compatibility with the english version by a group of people who converted it back to english and compared the converted versions. The questionnaire consists of three parts. The first part was about socio-demographic characteristics; the second part was about participants' knowledge about anesthesia; and the third part was about professionals' attitudes towards anesthesia. After informing each participant about the purpose of the study and obtaining informed consent, data collection began. After the questionnaires were filled out by the participants, the two trained data collectors compiled and checked the data for any conflicts that may have occurred during the data collection.

The development and translation of the questionnaire was the most challenging task, and it was developed by both the anesthetists and anesthesiologists. The questionnaire was pre-tested on 25 randomly selected health professionals. After pre-testing, some questions were modified to make them more understandable.

Attitude-related questions were answered as strongly agree, agree, disagree, strongly disagree, and none. the investigators prepared a total of 15 knowledge-related questions, of them 10 were closed-ended and could be scored objectively.

ELIGIBILITY:
Inclusion Criteria:

* All health professionals in Dessie comprehensive specialized hospital who are voluntary to participate in the study.

Exclusion Criteria:

1. Group who are not voluntary,
2. Anesthetists/anesthesiologists
3. other institution medical staff worked as a contract at Dessie hospital

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: the population of this study was all medical staff working at Dessie referral hospital. this staff includes all specialties like Nursing, laboratory, midwifery, medical doctors, psychiatry nurses, radiology, and others. all have the chance to participation
Sampling Method: Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
To determine health professionals' knowledge on anesthesia service | from may 1 to septamber 30 2022
  The knowledge outcome was measured by dividing the correct answer to the total questions(15) as a percentage. Percentage scores <50% are poor, 50%-75% moderate, and >75% good.
To determine health professionals' attitude on anesthesia service | from may 1 to septamber 30 2022
  The attitude was measured by the Likert scale as agree, strongly agree, disagree, strongly disagree, or none. The likert scale is used to measure the percentage of positive or negative attitudes toward certain issues. Agree and strongly agree are considered as relatively similar responses while disagree and strongly disagree as similar responses. . Percentage scores <50% are poor, 50%-75% moderate, and >75% good.

CONTACTS AND LOCATIONS:
Overall Officials: Woldemichael, Principal Investigator — Wollo Universty
Locations (1):
- Dessie comprehensive specilized hospital, Dessie, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No